CLINICAL TRIAL: NCT00855309
Title: Low Dose Versus Weight-based Intravenous Acyclovir for Herpes Simplex Virus Prophylaxis in the Neutropenic Patient
Brief Title: Acyclovir in Preventing Herpes Simplex Virus Infection in Patients With Neutropenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00007690; P30CA012197 (NIH); CCCWFU-98608; IRB00007690
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Herpes Simplex
Keywords: chemotherapeutic agent toxicity; renal toxicity; infection; neutropenia
MeSH Terms: conditions — Herpes Simplex; Infections; Neutropenia | interventions — Acyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Patients receive weight-based IV acyclovir sodium every 8 or 12 hours.
  Interventions: Drug: acyclovir sodium
- Arm II (Experimental): Patients receive low-dose IV acyclovir sodium every 8 or 12 hours.
  Interventions: Drug: acyclovir sodium

INTERVENTIONS:
Drug: acyclovir sodium — Given IV

SUMMARY:
RATIONALE: Acyclovir may be effective in preventing herpes simplex virus infection in patients with neutropenia.

PURPOSE: This randomized phase III trial is studying the side effects of acyclovir and is comparing two doses of acyclovir in preventing herpes simplex virus infection in patients with neutropenia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the difference in nephrotoxicity between low-dose and weight-based intravenous acyclovir sodium as herpes simplex virus infection prophylaxis in patients with neutropenia.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive weight-based IV acyclovir sodium every 8 or 12 hours.
* Arm II: Patients receive low-dose IV acyclovir sodium every 8 or 12 hours. Treatment continues for approximately 2 weeks unless clinical herpes simplex virus infection is confirmed or the patient is no longer neutropenic.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older.
* Receiving treatment in inpatient oncology services at Wake Forest University Baptist Medical Center
* Receiving chemotherapy or have received chemotherapy within the past 2 weeks
* Seropositive herpes simplex virus (HSV)-1 or HSV-2 immunoglobulin antibody assay
* Creatinine clearance ≥ 50 mL/min
* Intravenous acyclovir sodium therapy is deemed necessary by the physician based upon clinical judgement (i.e., mucositis, vomiting, decreased GI absorption)

Exclusion Criteria:

* Pregnant or nursing
* Hypersensitivity to acyclovir sodium
* High tumor burden (i.e., WBC > 50,000/mm^3 at admission)
* Neutropenic, defined as one of the following:
* ANC < 500/mm^3
* ANC < 1,000/mm^3 with a predicted decrease to 500/mm^3
* Active HSV infection, as evidenced by any of the following:
* Positive HSV cultures
* Oral lesions
* Receiving 5 mg/kg acyclovir sodium every 8 hours

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2008-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Jay Brown, PharmD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Weight-based IV Acyclovir: Patients receive weight-based IV acyclovir sodium every 8 or 12 hours.
- Low-dose IV Acyclovir: Patients receive low-dose IV acyclovir sodium every 8 or 12 hours.
Period: Overall Study
Arm/Group | Weight-based IV Acyclovir | Low-dose IV Acyclovir
Started | 57 | 55
Completed | 56 | 55
Not Completed | 1 | 0
Not completed — patient never recieved drug | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 57 | 55 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 39 | 81
  >=65 years | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (13.5) | 53.3 (14.4) | 54.4 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 27 | 51
  Male | 33 | 28 | 61
Region of Enrollment [Number; unit: participants]
  United States | 57 | 55 | 112

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Incidence of Nephrotoxicity, Defined as a Serum Creatinine ≥ 2 Times the Patient's Baseline
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 56 | 55
participants | 2 | 3

ADVERSE EVENTS:
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/55
Other Adverse Events (participants affected / at risk) | 2/56 | 3/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=56) | Arm II (N=55)
Nephrotoxicity (Renal and urinary disorders) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
per the protocol, only nephrotoxicities (as measured by Creatinine increase over baseline were observed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes